CLINICAL TRIAL: NCT04290130
Title: Dynamic Neural Mechanisms of Audiovisual Speech Perception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Columbia University (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael Beauchamp, PhD, Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 844668
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Speech Perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of brain activity using electrodes. — We will present audiovisual speech and record neural responses.

SUMMARY:
Understanding speech is one of the most important functions of the human brain. We use information from both the auditory modality (the voice the of person we are talking to) and the visual modality (the facial movements of the person we are talking to) to understand speech. We will use intracranial encephalography to study the organization and operation of the brain during audiovisual speech perception.

ELIGIBILITY:
Inclusion Criteria:

* must be undergoing neurosurgery for the treatment of a brain disorder

Exclusion Criteria:

* must have corrected-to-normal vision and hearing

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of neural activity | During the procedure.
  The name of the measurement is the broadband high-frequency activity (BHA) in the brain in response to audiovisual speech. The unit of measure is % increase in power from pre-stimulus baseline. The name of the measurement tool is intracranial EEG, recordings of the raw voltage signal from each electrode implanted in the brain. The voltage-by-time signal will be converted to spectral space using a wavelet transform, and the magnitude of the power between 70 and 150 Hz inclusive in a time window between 0 ms and 500 ms after stimulus onset will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No